CLINICAL TRIAL: NCT00904319
Title: Optimizing Mobility in Older Adults With Knee Osteoarthritis: Aquatic Power Training
Brief Title: Aquatic Power Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Neil A. Segal, MD, The University of Iowa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200903762
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee pain; power training; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aquatic (Experimental): Aquatic Power Training
  Interventions: Other: Aquatic Power Training

INTERVENTIONS:
Other: Aquatic Power Training — Aquatic power training program with an exercise specialist 2/week for 6 weeks.

SUMMARY:
Knee Osteoarthritis (OA) accounts for a significant proportion of mobility limitations and is one of the most disabling problems facing the growing population of older adults. The purpose of this research is to reduce disablement of older adults with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
Aquatic based training can offer many of the same benefits associated with a land based exercises but water has certain properties that provide a more gentle and welcoming environment for exercising. Buoyancy in water counteracts gravity to support the weight of the subject and decrease the forces put on the joints. Viscosity of water can provide resistance proportional to the effort exerted and with gentle friction enhancing proprioceptive feedback. Immersing in warm water can cause an increase in body temperature due to specific heat and thermal conductivity, which can cause blood vessels to dilate. In addition, hydrostatic forces reduce edema, increasing venous return and healthy circulation. [Prins, 1999]; [Wilder, 1998]

Studies have shown that water based exercise has been proven to significantly decrease pain in people with knee osteoarthritis compared to those in a land based exercise program. [Silva, 2003] In comparing an aquatic physical therapy session to a no intervention group the aquatic program resulted in less pain, improved physical function, quality of life, and strength. [Hinman, 2007]

The purpose of this research study is to determine whether an aquatic therapy program aimed at increasing muscle power will be effective in improving knee symptoms and mobility in men and women with symptomatic knee osteoarthritis.

The purpose of this study is to assess the efficacy of aquatic power training for improving mobility limitations, disability and quality of life in older adults with symptomatic knee OA.

Hypothesis 1: In older adults with symptomatic knee OA, a 6-week aquatic power training intervention will reduce lower limb mobility limitations (400m walk time).

Hypothesis 2: In comparison to baseline measures, at 6-week follow-up, there will be improvements in a) lower limb function (LLFDI), b) quality of life (KOOS Knee QOL),c) knee OA specific pain (KOOS pain) scores, and d) vastus lateralis muscle bulk (thigh muscle). These changes will be sustained at 12 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Symptomatic knee osteoarthritis (knee osteoarthritis diagnosed by the American College of Rheumatology criteria and frequent knee symptoms)

Exclusion Criteria:

* bilateral knee replacement
* acute or terminal illness
* unstable cardiovascular condition or other medical conditions that may impair ability to participate such as pulmonary disease requiring use of supplement oxygen, or lower limb musculoskeletal surgery in the past 6 months
* unwilling to be in a pool (approximately 4 feet deep)
* 400m walk time equal to or slower than the median for sex and decade:

M 50's 250.2 60's 289.9 70's+ 290.8

F 50's 315.9 60's 305.2 70's+ 292.5

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
400 meter walk time | 0, 6, and 12 weeks

SECONDARY OUTCOMES:
Lower limb function (LLFDI) | 0, 6, and 12 weeks
Quality of life (KOOS) | 0, 6, and 12 weeks
Knee osteoarthritis pain (KOOS pain scores) | 0 and 6 weeks
Vastus lateralis muscle bulk | 0, 2, 6, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States